CLINICAL TRIAL: NCT01310829
Title: Developing Providers' Communication and Counseling Skills in Cancer Genetics Using Virtual Reality
Brief Title: Virtual Reality Intervention in Cancer Genetics
Status: Withdrawn | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0456
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Cancer; Prevention Harmful Effects
Keywords: Genetic counselor; Genetic counseling degree program; Genetic counseling students; Virtual reality-based intervention; VR; Genetic counseling; hereditary cancers; Questionnaires; Physiological measurements; Skin sensors
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Virtual Reality: Board-eligible or board-certified genetic counselors and students evaluate a virtual reality-based intervention using questionnaires and physiological measurements.
  Interventions: Behavioral: Questionnaires; Behavioral: Physiological Measurements; Behavioral: Virtual Reality Scene Viewing

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires completed before and after viewing virtual reality scenes, taking about 30 minutes to complete.
  Other Names: Survey
Behavioral: Physiological Measurements — Small sensors applied to skin will measure heart rate and sweat amounts while participants view a virtual reality scene.
Behavioral: Virtual Reality Scene Viewing — Prototype virtual reality application that demonstrates a provider-patient communication scenario commonly encountered in genetic counseling for hereditary cancers.
  Other Names: VR technology

SUMMARY:
The goal of this study is to evaluate a virtual reality-based intervention for training health care providers who are not genetics specialists to effectively communicate with and counsel patients regarding cancer genetics.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete questionnaires, have your physiological measurements recorded, and view virtual reality scenes.

Questionnaires:

You will fill out questionnaires before and after viewing the virtual reality scenes. Before viewing the virtual reality scenes, you will answer questions about your demographic, educational and professional background and about the likelihood of becoming engaged in a virtual environment. After viewing the virtual reality scenes, you will answer questions to evaluate the scenes. You also will be asked to provide additional comments about the virtual reality scenes during a brief interview. In total, these questionnaires should take about 30 minutes total to complete.

Physiological Measurements:

Your heart rate and the amount you sweat will be recorded during the virtual reality scene (described below) by applying small sensors to your skin.

After you have completed the first set of questionnaires, you will sit in a recliner and the sensors will be placed on your rib cage and hand. The sensors that measure heart rate will be placed in the following locations: your lower left rib cage, just under your right collar bone, and just under your left collar bone. The sensors that measure the amount you sweat will be placed on the palm of your hand.

The Virtual Reality Scenes:

You will sit in a recliner and be asked to put on a virtual reality helmet, which has goggles and noise-cancelling headphones. You will be told how to wear the helmet and use the hand-held controller.

You will first view a sample virtual reality scene to help orient you to the technology. The experience of virtual reality may involve multiple senses. For example, you may hear, smell, and feel sensations (such as mild vibrations) that are associated with the scenes you are viewing.

After you become comfortable using the technology, you will view a virtual reality scenario that depicts a typical session in cancer genetic counseling. The scenario will depict a virtual patient who is being seen for genetic counseling. You will be encouraged to speak to and interact with the virtual patient as you would with a real patient. The interaction with the virtual patient will be recorded. It is estimated that you will spend about 30 minutes in the genetic counseling scene with the virtual patient.

After the scene has ended, the equipment and sensors will be removed, and you will be asked to complete the second set of questionnaires and the brief interview.

It is expected that it will take up to 2 hours to complete all study procedures.

This is an investigational study.

Up to 21 people will take part in this study at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Genetic counselors: Board-eligible or board-certified genetic counselor
2. Genetic counseling students: Currently enrolled and in good standing in an accredited genetic counseling degree program
3. 18 years of age or older

Exclusion Criteria:

1. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Genetic counselors and genetic counseling students
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Proof of concept for Virtual Reality (VR) Technology as Training Method About Hereditary cancer risk and genetic testing | 2 hours
  Proof of concept for VR application established if VR prototype successfully evokes a sense of presence and co-presence (measured by the PQ and CPQ questionnaires, respectively). Responses to the PQ and CPQ given on a 7-point scale, with higher scores indicating higher degrees of presence and co-presence where mean scores above 4 considered high degree of presence and co-presence.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PHD, MPH, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org